CLINICAL TRIAL: NCT00557505
Title: A Phase 1 Pharmacokinetic And Pharmacodynamic Study Of PF-03732010 In Patients With Advanced Solid Tumors
Brief Title: A Study Of PF-03732010 In Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A9301001
Record Dates: First submitted 2007-11-12; First posted 2007-11-14 (Estimated); Results first posted 2012-03-26 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-02

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — PF-03732010 monoclonal antibody

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PF-03732010 (Experimental): Single Arm study
  Interventions: Drug: PF-03732010

INTERVENTIONS:
Drug: PF-03732010 — IV infusion. Escalating dose levels, starting at 0.5 mg/kg to Maximum Tolerated Dose. Cycle length of 4 weeks for first cycle, and 2 weekly for subsequently cycles was originally explored, yet based on emerging PK data the Cycle 1 duration is 2 weeks and then weekly. Number of Cycles: Until Progression or unacceptable toxicity develops.

SUMMARY:
P-cadherin may play a part in tumor growth; PF-03732010 is a new drug that inhibits P-cadherin. This study will test how well the drug is tolerated, and what effects there might be. Blood will also be taken to measure the amount of drug in blood.

ELIGIBILITY:
Inclusion Criteria:

* Advanced solid tumors refractory to (or intolerant of) established therapy known to provide clinical benefit, or for which there is no standard therapy
* Age >= 18 years of age
* Adequate bone marrow function as defined by: absolute neutrophil count (ANC) ≥1500/uL, hemoglobin ≥ 9 g/dL, platelets > 100,000/uL
* Adequate liver function as defined by: bilirubin < 1.5 x ULN, AST, ALT and ALP < 2.5 x ULN, or < 5 x ULN with documented liver and/or bone metastases
* Serum creatinine < 1.5 x ULN
* ECOG status 0-1
* Availability of biopsy tumor tissue (or fine needle aspirate) for testing of P-cadherin expression
* Tumor tissue (or fine needle aspirate) showing over-expression of P-cadherin
* Must be able to give written informed consent
* Be able to comply with scheduled study visits, treatment plans, laboratory tests and other procedures

Exclusion Criteria:

* Chemotherapy, radiotherapy, or any investigational cancer therapy within 4 weeks of study entry
* Patients with carcinomatous meningitis or untreated brain metastases.
* History of significant low platelet count, and/or bleeding disorders, requiring medical or surgical intervention
* History of significant bleeding episodes within 6 months, unless the source of bleeding has been resected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2007-12; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- Pfizer Investigational Site, Philadelphia, Pennsylvania, United States
- Pfizer Investigational Site, Parkville, Victoria, Australia
- Pfizer Investigational Site, Seoul, South Korea

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9301001&StudyName=A%20Study%20Of%20PF-03732010%20In%20Patients%20With%20Advanced%20Solid%20Tumors

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-03732010 0.5 mg/kg Biweekly: PF-03732010 infusion 0.5 milligram per kilogram (mg/kg) intravenously (IV) administered over 1 hour (hr) on Day 1 of cycle 1 (28 days cycle) and subsequently on Day 1 of each cycle (dosing interval of 14 days).
- PF-03732010 1.0 mg/kg Biweekly: PF-03732010 infusion 1.0 mg/kg IV administered over 1 hr on Day 1 of cycle 1 (28 days cycle) and subsequently on Day 1 of each cycle (dosing interval of 14 days).
- PF-3732010 2.0 mg/kg Biweekly: PF-03732010 infusion 2.0 mg/kg IV administered over 1 hr on Day 1 of cycle 1 (28 days cycle) and subsequently on Day 1 of each cycle (dosing interval of 14 days).
- PF-03732010 4.0 mg/kg Biweekly: PF-03732010 infusion 4.0 mg/kg IV administered over 1 hr on Day 1 of cycle 1 (28 days cycle) and subsequently on Day 1 of each cycle (dosing interval of 14 days).
- PF-03732010 8.0 mg/kg Biweekly: PF-03732010 infusion 8.0 mg/kg IV administered over 1 hr on Day 1 of cycle 1 (28 days cycle) and subsequently on Day 1 of each cycle (dosing interval of 14 days).
- PF-03732010 15.0 mg/kg Biweekly: PF-03732010 infusion 15.0 mg/kg IV administered over 1 hr on Day 1 of cycle 1 (28 days cycle) and subsequently on Day 1 of each cycle (dosing interval of 14 days).
- PF-03732010 4.0 mg/kg Weekly: PF-03732010 infusion 4.0 mg/kg IV administered over 1 hr on Day 1 of cycle 1 (14 days cycle) and subsequently on Day 1 of each cycle (dosing interval of 7 days).
- PF-03732010 8.0 mg/kg Weekly: PF-03732010 infusion 8.0 mg/kg IV administered over 1 hr on Day 1 of cycle 1 (14 days cycle) and subsequently on Day 1 of each cycle (dosing interval of 7 days).
- PF-03732010 15.0 mg/kg Weekly: PF-03732010 infusion 15.0 mg/kg IV administered over 1 hr on Day 1 of cycle 1 (14 days cycle) and subsequently on Day 1 of each cycle (dosing interval of 7 days).
Period: Overall Study
Arm/Group | PF-03732010 0.5 mg/kg Biweekly | PF-03732010 1.0 mg/kg Biweekly | PF-3732010 2.0 mg/kg Biweekly | PF-03732010 4.0 mg/kg Biweekly | PF-03732010 8.0 mg/kg Biweekly | PF-03732010 15.0 mg/kg Biweekly | PF-03732010 4.0 mg/kg Weekly | PF-03732010 8.0 mg/kg Weekly | PF-03732010 15.0 mg/kg Weekly
Started | 3 | 3 | 4 | 3 | 2 | 3 | 3 | 5 | 17
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 4 | 3 | 2 | 3 | 3 | 5 | 17
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Global deterioration of health | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Objective progression or relapse | 2 | 3 | 3 | 2 | 2 | 3 | 2 | 5 | 15
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- PF-03732010 0.5 mg/kg Biweekly: PF-03732010 infusion 0.5 mg/kg IV administered over 1 hr on Day 1 of cycle 1 (28 days cycle) and subsequently on Day 1 of each cycle (dosing interval of 14 days).
- Total: Total of all reporting groups
Arm/Group | PF-03732010 0.5 mg/kg Biweekly | PF-03732010 1.0 mg/kg Biweekly | PF-3732010 2.0 mg/kg Biweekly | PF-03732010 4.0 mg/kg Biweekly | PF-03732010 8.0 mg/kg Biweekly | PF-03732010 15.0 mg/kg Biweekly | PF-03732010 4.0 mg/kg Weekly | PF-03732010 8.0 mg/kg Weekly | PF-03732010 15.0 mg/kg Weekly | Total
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 2 | 3 | 3 | 5 | 17 | 43
Age, Customized [Number; unit: participants]
  18 to 44 years | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 5
  45 to 64 years | 1 | 1 | 3 | 2 | 2 | 1 | 1 | 3 | 13 | 27
  Equal to or greater than 65 years | 2 | 1 | 1 | 0 | 0 | 1 | 2 | 1 | 3 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 2 | 7 | 17
  Male | 2 | 1 | 3 | 2 | 1 | 2 | 2 | 3 | 10 | 26

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Time Frame: Baseline up to end of treatment (EOT) or withdrawal assessed up to Day 7 of last cycle
Population: MTD analysis population included all participants enrolled in the dose escalation part of the study who received at least 1 dose of study medication.
Measure: Number; unit: mg/kg
Arm/Group | PF-03732010 0.5 mg/kg Biweekly | PF-03732010 1.0 mg/kg Biweekly | PF-3732010 2.0 mg/kg Biweekly | PF-03732010 4.0 mg/kg Biweekly | PF-03732010 8.0 mg/kg Biweekly | PF-03732010 15.0 mg/kg Biweekly | PF-03732010 4.0 mg/kg Weekly | PF-03732010 8.0 mg/kg Weekly | PF-03732010 15.0 mg/kg Weekly
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 2 | 3 | 3 | 5 | 17
mg/kg | NA — MTD was not achieved since no participant experienced dose-limiting toxicity. | NA — MTD was not achieved since no participant experienced dose-limiting toxicity. | NA — MTD was not achieved since no participant experienced dose-limiting toxicity. | NA — MTD was not achieved since no participant experienced dose-limiting toxicity. | NA — MTD was not achieved since no participant experienced dose-limiting toxicity. | NA — MTD was not determined since schedule of administration of PF-03732010 was modified and so, the cohort was not expanded for determination of MTD. | NA — MTD was not achieved since no participant experienced dose-limiting toxicity. | NA — MTD was not achieved since only 1 participant experienced dose-limiting toxicity but none experienced dose-limiting toxicity at the next higher dose. | NA — MTD was not pursued since PF-03732010 serum concentration, attained after the dose of 15mg/Kg weekly, was above the projected efficacious trough concentration for at least 200 hrs.

2. Primary Outcome: Recommended Phase-2 Dose (RP2D)
Time Frame: Baseline up to EOT or withdrawal assessed up to Day 7 of last cycle
Population: Data was not analyzed, as development of the compound was terminated.
Measure: Number; unit: mg/kg
Arm/Group | PF-03732010 0.5 mg/kg Biweekly | PF-03732010 1.0 mg/kg Biweekly | PF-3732010 2.0 mg/kg Biweekly | PF-03732010 4.0 mg/kg Biweekly | PF-03732010 8.0 mg/kg Biweekly | PF-03732010 15.0 mg/kg Biweekly | PF-03732010 4.0 mg/kg Weekly | PF-03732010 8.0 mg/kg Weekly | PF-03732010 15.0 mg/kg Weekly
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-28 Day)]
Description: AUC (0-28 day)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-28 day).
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 5, 10, 24 hrs after the start of infusion of first dose, Day 3, 5, 8, 11 of cycle 1; pre-dose and 1 hr after start of infusion in every other cycle starting from cycle 2 up to Week 4, 8 and 12 after last dose or withdrawal
Population: Data was not summarized, as development of the compound was terminated.
Measure: Geometric Mean (Standard Deviation); unit: nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | PF-03732010 0.5 mg/kg Biweekly | PF-03732010 1.0 mg/kg Biweekly | PF-3732010 2.0 mg/kg Biweekly | PF-03732010 4.0 mg/kg Biweekly | PF-03732010 8.0 mg/kg Biweekly | PF-03732010 15.0 mg/kg Biweekly
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax)
Time Frame: as for outcome 3
Population: Data was not summarized, as development of the compound was terminated.
Measure: Median (Full Range); unit: hr
Arm/Group | PF-03732010 0.5 mg/kg Biweekly | PF-03732010 1.0 mg/kg Biweekly | PF-3732010 2.0 mg/kg Biweekly | PF-03732010 4.0 mg/kg Biweekly | PF-03732010 8.0 mg/kg Biweekly | PF-03732010 15.0 mg/kg Biweekly | PF-03732010 4.0 mg/kg Weekly | PF-03732010 8.0 mg/kg Weekly | PF-03732010 15.0 mg/kg Weekly
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Minimum Observed Serum Trough Concentration (Cmin)
Time Frame: as for outcome 3
Population: Data was not summarized, as development of the compound was terminated.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-03732010 0.5 mg/kg Biweekly | PF-03732010 1.0 mg/kg Biweekly | PF-3732010 2.0 mg/kg Biweekly | PF-03732010 4.0 mg/kg Biweekly | PF-03732010 8.0 mg/kg Biweekly | PF-03732010 15.0 mg/kg Biweekly | PF-03732010 4.0 mg/kg Weekly | PF-03732010 8.0 mg/kg Weekly | PF-03732010 15.0 mg/kg Weekly
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Maximum Observed Serum Concentration (Cmax)
Time Frame: as for outcome 3
Population: Data was not summarized, as development of the compound was terminated.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-03732010 0.5 mg/kg Biweekly | PF-03732010 1.0 mg/kg Biweekly | PF-3732010 2.0 mg/kg Biweekly | PF-03732010 4.0 mg/kg Biweekly | PF-03732010 8.0 mg/kg Biweekly | PF-03732010 15.0 mg/kg Biweekly | PF-03732010 4.0 mg/kg Weekly | PF-03732010 8.0 mg/kg Weekly | PF-03732010 15.0 mg/kg Weekly
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-14 Day)]
Description: AUC (0-14)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-14 day).
Time Frame: as for outcome 3
Population: Data was not summarized, as development of the compound was terminated.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | PF-03732010 4.0 mg/kg Weekly | PF-03732010 8.0 mg/kg Weekly | PF-03732010 15.0 mg/kg Weekly
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast).
Time Frame: as for outcome 3
Population: Data was not summarized, as development of the compound was terminated.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | PF-03732010 0.5 mg/kg Biweekly | PF-03732010 1.0 mg/kg Biweekly | PF-3732010 2.0 mg/kg Biweekly | PF-03732010 4.0 mg/kg Biweekly | PF-03732010 8.0 mg/kg Biweekly | PF-03732010 15.0 mg/kg Biweekly | PF-03732010 4.0 mg/kg Weekly | PF-03732010 8.0 mg/kg Weekly | PF-03732010 15.0 mg/kg Weekly
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Clearance (CL)
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: as for outcome 3
Population: Data was not summarized, as development of the compound was terminated.
Measure: Geometric Mean (Standard Deviation); unit: Liter/hr
Arm/Group | PF-03732010 0.5 mg/kg Biweekly | PF-03732010 1.0 mg/kg Biweekly | PF-3732010 2.0 mg/kg Biweekly | PF-03732010 4.0 mg/kg Biweekly | PF-03732010 8.0 mg/kg Biweekly | PF-03732010 15.0 mg/kg Biweekly | PF-03732010 4.0 mg/kg Weekly | PF-03732010 8.0 mg/kg Weekly | PF-03732010 15.0 mg/kg Weekly
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Apparent Volume of Distribution (Vd)
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug.
Time Frame: as for outcome 3
Population: Data was not summarized, as development of the compound was terminated.
Measure: Geometric Mean (Standard Deviation); unit: Liter
Arm/Group | PF-03732010 0.5 mg/kg Biweekly | PF-03732010 1.0 mg/kg Biweekly | PF-3732010 2.0 mg/kg Biweekly | PF-03732010 4.0 mg/kg Biweekly | PF-03732010 8.0 mg/kg Biweekly | PF-03732010 15.0 mg/kg Biweekly | PF-03732010 4.0 mg/kg Weekly | PF-03732010 8.0 mg/kg Weekly | PF-03732010 15.0 mg/kg Weekly
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Objective Response of Complete Response or Partial Response
Description: Number of participants with objective response based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). CR are those that persist on repeat imaging study at least 4 weeks after initial documentation of response. PR are those with at least 30 percent decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: Baseline to disease progression or 4 weeks after the first dose and then every 6 weeks up to Week 37
Population: Data was not analyzed, as antitumor activity was not observed.
Measure: Number; unit: participants
Arm/Group | PF-03732010 0.5 mg/kg Biweekly | PF-03732010 1.0 mg/kg Biweekly | PF-3732010 2.0 mg/kg Biweekly | PF-03732010 4.0 mg/kg Biweekly | PF-03732010 8.0 mg/kg Biweekly | PF-03732010 15.0 mg/kg Biweekly | PF-03732010 4.0 mg/kg Weekly | PF-03732010 8.0 mg/kg Weekly | PF-03732010 15.0 mg/kg Weekly
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Other Pre Specified Outcome: Human Anti-Human Antibody (HAHA) Levels
Description: HAHA are indicators of immunogenicity to PF-03732010.
Time Frame: Pre-dose on Day 1 of Cycle 2 and Day 1 of every other cycle up to Week 4, 8 and 12 after the last dose or withdrawal
Population: Data was not analyzed, as development of the compound was terminated.
Measure: Mean (Standard Deviation); unit: microgram/mL
Arm/Group | PF-03732010 0.5 mg/kg Biweekly | PF-03732010 1.0 mg/kg Biweekly | PF-3732010 2.0 mg/kg Biweekly | PF-03732010 4.0 mg/kg Biweekly | PF-03732010 8.0 mg/kg Biweekly | PF-03732010 15.0 mg/kg Biweekly | PF-03732010 4.0 mg/kg Weekly | PF-03732010 8.0 mg/kg Weekly | PF-03732010 15.0 mg/kg Weekly
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Other Pre Specified Outcome: Change From Baseline in Standardized Uptake Values (SUV) of 18F-fluoro-3'-Deoxy-3'-L-fluorothymidine Positron Emission Tomography (FLT-PET)
Time Frame: Baseline, cycle 3 and after 8 weeks
Population: Data was not analyzed, as development of the compound was terminated.
Measure: Mean (Standard Deviation); unit: standardized uptake value (SUV)
Arm/Group | PF-03732010 0.5 mg/kg Biweekly | PF-03732010 1.0 mg/kg Biweekly | PF-3732010 2.0 mg/kg Biweekly | PF-03732010 4.0 mg/kg Biweekly | PF-03732010 8.0 mg/kg Biweekly | PF-03732010 15.0 mg/kg Biweekly | PF-03732010 4.0 mg/kg Weekly | PF-03732010 8.0 mg/kg Weekly | PF-03732010 15.0 mg/kg Weekly
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Other Pre Specified Outcome: Time to Disease Progression
Description: Time in weeks from start of study treatment to first documentation of objective disease progression or death due to disease, whichever comes first.
Time Frame: Baseline to disease progression or 4 weeks after the first dose and then every 6 weeks up to Week 37
Population: Data was not analyzed, as antitumor activity was not observed.
Measure: Median (Full Range); unit: weeks
Arm/Group | PF-03732010 0.5 mg/kg Biweekly | PF-03732010 1.0 mg/kg Biweekly | PF-3732010 2.0 mg/kg Biweekly | PF-03732010 4.0 mg/kg Biweekly | PF-03732010 8.0 mg/kg Biweekly | PF-03732010 15.0 mg/kg Biweekly | PF-03732010 4.0 mg/kg Weekly | PF-03732010 8.0 mg/kg Weekly | PF-03732010 15.0 mg/kg Weekly
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

15. Other Pre Specified Outcome: Change From Baseline in Circulating Tumor Cells (CTC) Concentration in Blood
Time Frame: Pre-dose (baseline), Day 8 cycle 1, Day 1 Cycle 2 and Day 1 of every other cycle starting from cycle 3 up to EOT or withdrawal
Population: Data was not analyzed, as development of the compound was terminated.
Measure: Number; unit: cells/mL
Arm/Group | PF-03732010 0.5 mg/kg Biweekly | PF-03732010 1.0 mg/kg Biweekly | PF-3732010 2.0 mg/kg Biweekly | PF-03732010 4.0 mg/kg Biweekly | PF-03732010 8.0 mg/kg Biweekly | PF-03732010 15.0 mg/kg Biweekly | PF-03732010 4.0 mg/kg Weekly | PF-03732010 8.0 mg/kg Weekly | PF-03732010 15.0 mg/kg Weekly
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

16. Other Pre Specified Outcome: Change From Baseline in Leucocyte Subtypes
Time Frame: Baseline, Day 1 cycle 1, Day 1 Cycle 2, Day 1 of every other cycle starting from cycle 3 up to EOT or withdrawal
Population: Data was not analyzed, as development of the compound was terminated.
Measure: Number; unit: cells/mL
Arm/Group | PF-03732010 0.5 mg/kg Biweekly | PF-03732010 1.0 mg/kg Biweekly | PF-3732010 2.0 mg/kg Biweekly | PF-03732010 4.0 mg/kg Biweekly | PF-03732010 8.0 mg/kg Biweekly | PF-03732010 15.0 mg/kg Biweekly | PF-03732010 4.0 mg/kg Weekly | PF-03732010 8.0 mg/kg Weekly | PF-03732010 15.0 mg/kg Weekly
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

17. Other Pre Specified Outcome: Change From Baseline in Cytokine Concentration
Time Frame: Pre-dose (baseline), 1, 6 and 24 hrs after start of infusion on Day 1 cycle 1
Population: Data was not analyzed, as development of the compound was terminated.
Measure: Mean (Standard Deviation); unit: picogram (pg)/mL
Arm/Group | PF-03732010 0.5 mg/kg Biweekly | PF-03732010 1.0 mg/kg Biweekly | PF-3732010 2.0 mg/kg Biweekly | PF-03732010 4.0 mg/kg Biweekly | PF-03732010 8.0 mg/kg Biweekly | PF-03732010 15.0 mg/kg Biweekly | PF-03732010 4.0 mg/kg Weekly | PF-03732010 8.0 mg/kg Weekly | PF-03732010 15.0 mg/kg Weekly
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

18. Other Pre Specified Outcome: Change From Baseline in Tumor Proteins Related to P-cadherin Signaling and/or Tumor Proliferation or Apoptosis by Immunohistochemistry (IHC)
Time Frame: Baseline and cycle 3
Population: Data was not analyzed, as development of the compound was terminated.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | PF-03732010 0.5 mg/kg Biweekly | PF-03732010 1.0 mg/kg Biweekly | PF-3732010 2.0 mg/kg Biweekly | PF-03732010 4.0 mg/kg Biweekly | PF-03732010 8.0 mg/kg Biweekly | PF-03732010 15.0 mg/kg Biweekly | PF-03732010 4.0 mg/kg Weekly | PF-03732010 8.0 mg/kg Weekly | PF-03732010 15.0 mg/kg Weekly
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | PF-03732010 0.5 mg/kg Biweekly | PF-03732010 1.0 mg/kg Biweekly | PF-3732010 2.0 mg/kg Biweekly | PF-03732010 4.0 mg/kg Biweekly | PF-03732010 8.0 mg/kg Biweekly | PF-03732010 15.0 mg/kg Biweekly | PF-03732010 4.0 mg/kg Weekly | PF-03732010 8.0 mg/kg Weekly | PF-03732010 15.0 mg/kg Weekly
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 2/4 | 0/3 | 0/2 | 1/3 | 1/3 | 0/5 | 4/17
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 4/4 | 3/3 | 2/2 | 3/3 | 3/3 | 5/5 | 13/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-03732010 0.5 mg/kg Biweekly (N=3) | PF-03732010 1.0 mg/kg Biweekly (N=3) | PF-3732010 2.0 mg/kg Biweekly (N=4) | PF-03732010 4.0 mg/kg Biweekly (N=3) | PF-03732010 8.0 mg/kg Biweekly (N=2) | PF-03732010 15.0 mg/kg Biweekly (N=3) | PF-03732010 4.0 mg/kg Weekly (N=3) | PF-03732010 8.0 mg/kg Weekly (N=5) | PF-03732010 15.0 mg/kg Weekly (N=17)
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Brain stem infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-03732010 0.5 mg/kg Biweekly (N=3) | PF-03732010 1.0 mg/kg Biweekly (N=3) | PF-3732010 2.0 mg/kg Biweekly (N=4) | PF-03732010 4.0 mg/kg Biweekly (N=3) | PF-03732010 8.0 mg/kg Biweekly (N=2) | PF-03732010 15.0 mg/kg Biweekly (N=3) | PF-03732010 4.0 mg/kg Weekly (N=3) | PF-03732010 8.0 mg/kg Weekly (N=5) | PF-03732010 15.0 mg/kg Weekly (N=17)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 5
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 2
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Saliva altered (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Tongue disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 1 | 1 | 2 | 1 | 0 | 2 | 3
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vaginal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 2
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue paralysis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Penile pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 1 | 0 | 0 | 1 | 2 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 1 | 0 | 1 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Haemorrhage (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Results are not provided because development of the study drug was terminated, as neither anti-tumor activity nor pharmacodynamic modulation was observed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.